CLINICAL TRIAL: NCT07204314
Title: A Randomized, Double-blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Once-Daily Oral Administration of Vortioxetine in Japanese Pediatric Patients 12 to 17 Years of Age With Major Depressive Disorder (MDD)
Brief Title: A Study of Vortioxetine in Japanese Pediatric Patients With Major Depressive Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vortioxetine-3023; U1111-1314-6051 (Other: WHO); jRCT2031250396 (Registry Identifier: jRCT)
Record Dates: First submitted 2025-09-30; First posted 2025-10-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vortioxetine (Experimental): Participants will receive the study drug, orally, once, daily (QD) for 14 weeks. The vortioxetine dose will be started at 10 mg per day, and can be increased to 20 mg per day.
  Interventions: Drug: Vortioxetine tablets
- Placebo (Placebo Comparator): Participants will receive the study drug, orally, once, daily (QD) for 14 weeks.
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Vortioxetine tablets — Vortioxetine tablets
  Other Names: Trintellix
  Arms: Vortioxetine
Drug: Placebo tablets — Placebo tablets
  Arms: Placebo

SUMMARY:
The main aim of the study is to check how well vortioxetine 10 mg/day or 20 mg/day works and to check for side effects compared to a placebo on depression symptoms in Japanese teenagers aged 12 to 17 years with a diagnosis of Major Depressive Disorder (MDD).

The overall time each participant will be in the study is about 20 weeks. This includes up to 15 days (about 2 weeks) to check who can take part, a 14-week period where everyone receives vortioxetine or a placebo, and after that, a 4-week period to check for any side effects after treatment.

During the study, participants will visit their clinic 13 times.

ELIGIBILITY:
Inclusion Criteria:

1. The Japanese participant is a male or female, aged 12 to 17 years at the time of informed consent (patients who turn 18 years during the trial will be allowed to continue in the trial).
2. The participant is capable of communicating with the site personnel.
3. The participant is able to understand the informed assent form or the ICF and parent(s)/legal guardian(s) are able to read and understand the ICF. The participant is able and willing to accept video recording at the assessment by the trial site and evaluation by third party evaluators (Central Evaluating Committee).
4. The participant has provided the written informed assent as much as possible to participation and parent(s)/legal guardian(s) signed the ICF.
5. The participant and parent(s)/legal guardian(s) are willing and able to attend trial appointments within the specified time windows.
6. The participant is an outpatient consulting a clinician.
7. The participant has a primary diagnosis of MDD or persistent depressive disorder and fully meet the criteria for major depressive episodes according to DSM-5-TR without psychotic features although co-morbid anxiety disorders will be permitted. The diagnoses will be confirmed using the MINI-KID.
8. The participant has a CDRS-R total score greater than or equal to 45 at the Screening Visit and at the Baseline A Visit (Week 0).
9. The participant has a CGI-S score greater than or equal to4 at the Screening Visit and at the Baseline A Visit (Week 0).
10. The participant has a PHQ-A score of greater than or equal to10 at the Baseline A Visit (Week 0).
11. The participant, if a female and is capable of producing viable ova, agrees to the following, for the period from the signing of ICF until 30 days after the last dose of trial intervention.

    * To use a highly effective or acceptable contraceptive method
    * To avoid donating ova
12. The participant, if a female, must have a confirmed negative urine pregnancy test at the Screening Visit

Exclusion Criteria:

1. The participant has previously been entered and moved to Phase A in this trial.
2. The participant has participated in a clinical trial less than 30 days before the Screening Visit.
3. The participant is a member of the trial personnel or of their immediate families or is a subordinate (or immediate family member of a subordinate) to any of the trial personnel.
4. The participant has been previously treated with vortioxetine.
5. The participant has the current or previous major depressive episode which was considered by the investigators to have been resistant to 2 or more adequate antidepressants treatments of at least 6-weeks duration each at sufficient doses.
6. The participant is under forced treatment.
7. The participant has experienced any environmental change (eg, hospitalization, change of residence) considered by the investigator to have the potential impact on the participant's disease situation or plans such environmental changes during the trial.
8. The participant is pregnant or breast-feeding.
9. The participant receives on-going psychotherapy (except for a supportive psychotherapy) that is started less than 3 months before the Baseline A Visit (Week 0) and/or that is planned to be intensified during the trial.
10. The participant has a history of severe drug allergy or hypersensitivity or known hypersensitivity to any of the IMPs or their excipients.
11. The participant has hereditary problems of fructose intolerance, glucose-galactose malabsorption, or sucrase-isomaltose insufficiency.
12. The participant has any current psychiatric disorder (DSM-5-TR criteria), including posttraumatic stress disorder (PTSD), obsessive-compulsive disorder (OCD), autism spectrum disorder (ASD), and attention-deficit/hyperactivity disorder (ADHD) established as the primary diagnosis, as assessed using the MINI-KID.
13. The participant has a medical history of substance use disorder (excluding nicotine, and caffeine) or alcohol use disorder (DSM-5-TR criteria) less than 6 months before the Screening Visit.
14. The participant has reported current use of or has tested positive for drugs of abuse (opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates, benzodiazepines, and cannabinoids, etc).
15. The participant suffers from medical, organic or drug cause mental disorders (DSM-5-TR criteria).
16. The participant has a known intellectual disability; or clinical evidence or known social or school history indicative of intellectual disability.
17. The participant has any other disorder for which the treatment takes priority over treatment of MDD or is likely to interfere with trial treatment or impair treatment compliance.
18. The participant has a history of moderate or severe head trauma; or other neurological disorders or systemic medical diseases that are, in the investigator's opinion, likely to affect central nervous system functioning.
19. The participant has a known first degree relative with a history of bipolar disorder.
20. The participant is unable to swallow tablets.
21. The participant has a history of cancer that has not been in remission for more than 5 years before the first dose of trial intervention.
22. The participant has or has had 1 or more of the following conditions that is/are considered clinically relevant in the context of the trial: neurological disorder, other psychiatric disorder, cardiovascular disease, seizure disorder or encephalopathy, congestive heart failure, cardiac hypertrophy, arrhythmia, bradycardia (pulse less than 50 bpm), respiratory disease, hepatic impairment or renal insufficiency, metabolic disorder, endocrinological disorder, gastrointestinal disorder, hematological disorder, infectious disorder, any clinically significant immunological condition, dermatological disorder, venereal disease, congenital or juvenile glaucoma or is at risk of acute narrow-angle glaucoma
23. The participant takes or has taken disallowed recent or concomitant medication, or it is anticipated that the participant will require treatment with at least one of the disallowed concomitant medications/procedures or treatment during the trial.
24. The participant has clinically significant abnormal vital signs at the Screening Visit.
25. The participant has 1 or more clinical laboratory test values outside the reference range, based on the blood and urine samples taken at the Screening Visit, which are of potential risk to the participant's safety; or the participant has, at the Screening Visit:

    * a serum creatinine value more than 1.5 times the upper limit of the reference range
    * a serum total bilirubin value more than 1.5 times the upper limit of the reference range
    * a serum ALT or AST value more than 2 times the upper limit of the reference range
26. The participant has an abnormal TSH level. Participant with thyroid disease may be enrolled in the trial provided they are stable and euthyroid at the discretion of the investigator.
27. The participant has, at the Screening Visit:

    * an abnormal ECG that is, in the investigator's opinion, clinically significant
    * a QTcF interval more than 450 ms (based on the Fridericia correction where QTcF = QT/RR0.33)
28. The participant has a disease or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the trial.
29. The participant is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.
30. The participant has attempted suicide within the last 12 months or is at significant risk of suicide (either in the opinion of the investigator or defined as a 'yes' to suicidal ideation questions 4 or 5 or answering 'yes' to suicidal behavior questions on the C-SSRS within the last 12 months).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Children Depression Rating Scale Revised version (CDRS-R) Total Score | Baseline, Week 14
  The CDRS-R is a clinician-rated scale to measure the severity of depression in children and adolescents. The CDRS-R is rated by a clinician following interviews with the child and parents/legal guardians and consists of 17 items out of which 3 items rate nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items are rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) are scored on a 5-point scale from 1 to 5. The total score ranges from 17 (normal) to 113 (severe depression). Higher scores indicate greater severity of depression.

SECONDARY OUTCOMES:
Change from Baseline in the CDRS-R Total Score at Each Time Point | Baseline, Week 2, 4, 6, 8, and 10
  The CDRS-R is a clinician-rated scale to measure the severity of depression in children and adolescents. The CDRS-R is rated by a clinician following interviews with the child and parents/legal guardians and consists of 17 items out of which 3 items rate nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items are rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) are scored on a 5-point scale from 1 to 5. The total score ranges from 17 (normal) to 113 (severe depression). Higher scores indicate greater severity of depression.
CDRS-R Response at Each Time Point | Week 2, 4, 6, 8, 10, and 14
  CDRS-R response is defined as at least 50 percent reduction in the CDRS-R total score from Baseline, calculated as the change from baseline divided by the result of subtracting 17 from the Baseline score. CDRS-R response at each time point will be reported.
Remission at Each Time Point | Week 2, 4, 6, 8, 10, and 14
  Remission is defined as less than or equal to 28 in the CDRS-R total score. Remission at each time point will be reported.
Change from Baseline in the Patient Health Questionnaire-9 for Adolescents (PHQ-A) at Each Time Point | Baseline, Week 4, 6 and 14
  The PHQ-A is a participant-rated scale designed to screen for depressive symptoms in adolescents. The 9 depression items are rated on a 4-point scale (0=Not at all; 1=Several days; 2=More than half the days; and 3=Nearly every day). The total score can range from 0 to 27, with higher scores indicating greater severity of depression.
Change from Baseline in the Digit Symbol Substitution Test (DSST) at Each Time Point | Baseline, Week 4 and 14
  The DSST is a paper-and-pencil cognitive test. After viewing a predetermined table of pairs of numbers and symbols, participants replace each symbol with its corresponding number, one by one. The number of correct symbols within the allowed time, usually 90 seconds, constitutes the score. The DSST score ranges from 0 to 133, with lower scores indicating lower cognitive function.
Change from Baseline in the Clinical Global Impression - Severity of Illness (CGI-S) Score at Each Time Point | Baseline, Week 2, 4, 6, 8, 10, and 14
  The CGI-S provides the clinician's impression of the participant's current state of mental illness. The clinician uses his or her clinical experience of this participant population to rate the severity of the participant's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill participants).
Score in the Clinical Global Impression - Global Improvement (CGI-I) at Each Time Point | Week 4, 6, 8, 10, and 14
  The CGI-I provides the clinician's impression of the participant's improvement (or worsening). The clinician assesses the participant's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Remission in the CGI-S Score at Each Time Point | Week 2, 4, 6, 8, 10, and 14
  Remission in the CGI-S score is defined as a CGI-S score of 1 or 2. Remission in the CGI-S score at each time point will be reported.
Response in the CGI-I Score at Each Time Point | Week 4, 6, 8, 10, and 14
  Response in the CGI-I Score is defined as defined as a CGI-I score of 1 or 2. Response in the CGI-I score at each time point will be reported.
Change from Baseline in the Sheehan Disability Scale - Adolescent Version (SDS-A) at Each Time Point | Baseline, Week 4 and 14
  The SDS-A assesses functional impairment in 3 major life domains: school/work, social life/leisure activities, and family life/home responsibilities. The 3 life domains are rated on a 11-point scale from 0 (Not at all) to 10 (Extremely). The total score ranges from 0 to 30, with higher scores indicating greater pathology.
Plasma Concentrations of Vortioxetine | Baseline, Week 6, 10, and 14

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (30):
- Japan (30):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Kaku Mental Clinic, Chūōku, Fukuoka
  - Jisenkai Nanko Psychiatric Institute, Shirakawa, Fukushima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - NHO Shikoku Medical Center for Children and Adults, Zentsujichó, Kagawa-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Tohoku University Hospital, Sendai, Miyagi
  - Miyakonojo Shinsei Hospital, Miyakonojō, Miyazaki
  - Nara Medical University Hospital, Kashihara, Nara
  - Bandai Mental Clinic, Chuo-ku, Niigata
  - University of the Ryukyus Hospital, Ginowan, Okinawa
  - Imurokokorono-clinic, Urasoe, Okinawa
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Harai Clinic, Chuo-ku, Tokyo
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Aiiku Clinic, Minato-ku, Tokyo
  - Pauroom, Minato-ku, Tokyo
  - Kai Kokoro Clinic, Suginome, Tokyo
  - Shin-Otsuka Clinic, Toshima-ku, Tokyo
  - Cerisier Heart Clinic, Kagoshima
  - Yuge Neuropsychiatric Hospital, Kumamoto
  - Chikama Clinic, Miyazaki
  - Osaka Metropolitan University Hospital, Osaka
  - Toyama University Hospital, Toyama

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/76775b052973403a